CLINICAL TRIAL: NCT06890559
Title: Enhancing Vaccination Uptake Through Points Redemption Based Financial Incentives and Digital Platforms: an Open-label Cluster Randomized Controlled Trial Utilizing Community Mobilization and Empowerment Strategies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Yan (Other)
Responsible Party: Sponsor-Investigator, Bo Yan, Doctor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZGL202502-6
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Vaccination Uptake
Keywords: financial incentive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- financial incentive group (Active Comparator)
  Interventions: Behavioral: financial incentive intervention based on a digital platform
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: financial incentive intervention based on a digital platform — The intervention will span a duration of 12 months. All residents in the 8 intervention subdistricts/townships are available for participation; each participant household needs to register a household account on the digital platform. Each family member who completes targeted vaccine uptake or related health behaviors can earn points through two point-recording routes. Reward points will be accumulated on a household basis to encourage family members' engagement. Points can be redeemed for gifts on the digital platform and are only valid once.
  Arms: financial incentive group

SUMMARY:
The overall goal is to develop and optimize a health digital platform and points redemption-based financial incentive interventions for the promotion of non-National Immunization Program (non-NIP) vaccination uptake and related preventative behaviors in China, and formulate a low-cost, labor-saving and replicable pattern. The primary objective is to develop and optimize a digital platform-based point-redemption and financial incentive system and evaluate the effectiveness of the interventions for improving non-NIP vaccines coverage and related preventive behaviors.The main questions it aims to answer are:

H1: Participants allocated to the intervention group will demonstrate a 3% increase in vaccine doses of targeted non-NIP vaccines, including HPV vaccines, influenza vaccines, pneumonia vaccines, rotavirus vaccines, varicella vaccines, and haemophilus Influenza Type B polysaccharide conjugate (Hib) vaccines, compared to those in the control group at the 12-month follow-up.

H2: Participants allocated to the intervention group will exhibit a 5% increase in the prevalence of related preventive behaviors compared to those in the control group at the 12-month follow-up.

Researchers will compare the financial incentive intervention to the routine activities to see if the intervention works to improve the vacciantion rate of non-NIP vaccines.

Participants will:

1. Participants can automatically input their health behaviors through the digital platform, and the back-end will verify the information with data provided by the township hospitals or community health centers.
2. A QR code will be implemented at each township hospital or community health center. Participants will scan the QR code after completing vaccination or other related preventive behaviors. The digital platform will automatically record points for each completed behavior.
3. Use accumulated points to redeem gifts on the system, including household goods, electronic products, and free or discounted health services.

ELIGIBILITY:
Inclusion Criteria:

* Do not move from the original research and implementation site within the next year;
* Voluntarily participate in the study and sign the informed consent;
* No mental disorder or cognitive impairment, able to understand and cooperate with research requirements.

Exclusion Criteria:

* Have contraindications related to vaccination;
* The state of the body during the intervention period is not suitable for vaccination.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The number of targeted non-NIP vaccine doses per 1,000 person-years | one year
  The primary outcome of interest is the number of targeted non-NIP vaccine doses per 1,000 person-years. The targeted vaccines in this study include HPV vaccines, influenza vaccines and pneumonia vaccines.

SECONDARY OUTCOMES:
Number of cervical cancer screenings, medical checkups for the elderly, and check-ups for children during the intervention period | one year
  Preventive behaviors related to vaccination, such as cervical cancer screening, medical checkups for the elderly,and check-ups for children during the intervention period. We will count the total number of occurrences through the participant's medical records and the number of times these behaviours are self-reported through the digital platform.

IPD SHARING:
Plan to Share IPD: No